CLINICAL TRIAL: NCT06825000
Title: The Effects of Science Education on Beliefs and Wellness
Brief Title: Scientific Information and Beliefs About Psychological Therapy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Golnaz Tabibnia, Assistant Research Psychologist, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3274
Record Dates: First submitted 2025-01-23; First posted 2025-02-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-02

CONDITIONS: Anxiety
Keywords: beliefs; mindsets; exposure therapy; neuroscience education; psycho-education; neuro-education
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuro-Ed Group (Experimental): neuroscience education
  Interventions: Behavioral: neuro-education
- Psycho-Ed Group (Active Comparator): psychological science education
  Interventions: Behavioral: psycho-education

INTERVENTIONS:
Behavioral: neuro-education — 30 minutes of videos about the neuroscience of stress, fear, emotion-regulation, and therapy.
  Other Names: neuroscience education; Neuro-Ed; NeuroEd
  Arms: Neuro-Ed Group
Behavioral: psycho-education — 30 minutes of videos about the psychological science of stress, fear, emotion-regulation, and therapy.
  Arms: Psycho-Ed Group

SUMMARY:
The success of psychological therapy can be impacted by patients' beliefs, such as their belief in their own ability to complete therapy and their belief that therapy will work. The goal of this clinical trial is to learn whether and when scientific information about distress and coping can affect beliefs about psychological therapy in adults who experience anxiety. This study will compare two different types of scientific information in a one-hour study. Participants will view educational videos for 30 minutes and complete surveys, including quiz questions about the videos and surveys about their beliefs about psychological therapy.

ELIGIBILITY:
Inclusion Criteria:

* Probable anxiety disorder based on the Overall Anxiety Severity and Impairment Scale (OASIS) score
* Fluent in English
* Willingness and ability to comply with the protocol
* Age 18-80
* The ability to enroll in the study through Prolific.com

Exclusion Criteria:

* Having previously seen the study's videos

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Treatment Self-Efficacy | Immediately before and immediately after watching the videos
  Measured through self-report on selected items from a version of the validated Bergen Genetic Counseling Self-Efficacy Scale that was previously adapted for treatment self-efficacy in anxiety disorders. The items are rated on a scale of 1-10, with higher numbers indicating greater self-efficacy.
Treatment Expectancy | Immediately before and immediately after watching the videos
  Measured through self-report on a subscale of the validated Credibility/Expectancy Questionnaire, assessing participants' expectation of treatment efficacy. Each item is rated on a scale of 1-9 or 0%-100%, with higher numbers indicating more optimistic expectancy.

SECONDARY OUTCOMES:
Treatment Acceptability | Immediately after watching the videos
  Participants will rate on a scale of 1-7 how useful, interesting, credible, and easy-to-understand they found the information in the videos. Greater numbers indicate greater acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Golnaz Tabibnia, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD that underlie results in a publication may be provided to qualified researchers with academic interest in science education and mental health. Approval of the request and execution of all applicable agreements may be prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data requests can be submitted starting 9 months after article publication, and the data will be made accessible for up to 5 years after study completion.
Access Criteria: Researchers requesting data will first be asked to provide a research proposal. Pending approval of the proposal, they will then be asked to sign a data sharing agreement, which will include restrictions against attempting to identify study participants, on redistribution of the data to third parties, on use of the data for commercial purposes, as well as requirements to electronically secure the data while in use, to destroy the data after analyses are completed, for reporting responsibilities, and for proper acknowledgement of the data resource.